CLINICAL TRIAL: NCT03178721
Title: Regulatory BCells in Systemic Lupus Erythematosus and Its Relation to Atherosclerosis and Disease Activity
Brief Title: Regulatory BCells in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Shawky, principle investegator, Assiut University
Other Study IDs: breg
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 1- 5ml fresh human peripheral whole blood was layered over a ficoll density gradient to isolate PBMCs. Breg cells will be sorted by fluorescently labelling PBMCs to identify Breg cells Quantification of the percentage of specific phenotype CD19+ CD38hi CD24hi of B-reg by using flow cytometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Systemic lupus erythematosus with atherosclerosis
  Interventions: Diagnostic Test: blood sample
- 2: Systemic lupus erythematosus without atherosclerosis
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — study B regulatory in blood and its correlation with atherosclerosis
  Other Names: Coronary calcium scoring: all participants will be scanned using a 64-slice CT scanner and Carotid intimae media thickness (CIMT): Carotid artery ultrasonography

SUMMARY:
Systemic lupus erythematosus , the archetypal multisystem autoimmune disease, presents many diagnostic and management challenges. One such challenge is the excess cardiovascular disease observed in patients with Systemic lupus erythematosus . Coronary heart disease and other manifestations of atherosclerosis continue to be a major cause of death in patients with Systemic lupus erythematosus.Regulatory B-cells have been identified as a negative regulator of the immune system that inhibit pathological immune response by suppressing both uncontrolled protective immune response and damaging autoimmune responses

DETAILED DESCRIPTION:
Regulatory B cells have been identified as an IL10 producing B cells subsets that are characterized by the expression of CD19 CD24hiCD38hi . Breg cells can inhibit inflammatory responses in autoimmune disease, like Systemic lupus erythematosus, via the production of IL-10 (an antiatherogenic cytokine) which will suppress TNF- α production by monocytes leading to inhibition of T cell-mediated inflammation. Regulatory B have a vital role in immune tolerance and their deficiency resulted in exacerbation of autoimmunity . Evidence suggests Breg in autoimmune disease may be dysfunctional .

In this proposal, We suggest IL-10 production by Breg confers an atheroprotective role. In Systemic lupus erythematosus, Regulatory B ability to control atherosclerosis is reduced therefore, we will test the hypothesis that Regulatory B play an important role in both autoimmunity and accelerated atherosclerosis and dysfunction in Regulatory B from autoimmune disease may or may not result in a reduced ability to control atherosclerosis .

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory Diagnosis of Systemic Lupus disease.
* Must be adult.

Exclusion Criteria:

* Patients with clinical atherosclerotic vascular disease
* pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult patients with systemic lupus erythematosus
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-25 (Estimated); Primary Completion 2018-06-25 (Estimated); Study Completion 2018-07-25 (Estimated)

PRIMARY OUTCOMES:
Coronary calcium scoring | 1year
  using Agatston score none (Agatston 0 U) mild (Agatston 1-99 U) moderate(Agatston 100-399 U) high(Agatston >400 U)

IPD SHARING:
Plan to Share IPD: No